CLINICAL TRIAL: NCT04584060
Title: Conventional VS Enhanced Recovery After Surgery Protocols in Emergency GIT Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Raouf Rida Naguib, Resident doctor, Assiut University
Other Study IDs: ERAS in emergency
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Patient Presented With Acute Abdomen; Patient Undergoing Urgent GIT Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional: Fatsing for at least 6 hours pre-operative, No restriction of IV fluids and traditional analgesia including opiates. Post-operative Ambulation-as per patients' own request, Removal of urinary catheter when patient ambulates, patient will keep fasting for 3 days postoperative, oral fluids for 3 days, semi-solid for another 3 days and then can take full diet, removal of nasogastric tube just before starting oral fluids, drain removal just before discharge.
- ERAS: Preoperative information, education and counselling, If possible, Clear fluids are allowed up to 2 h and solids up to 6 h prior to induction of anaesthesia, Short acting anesthetic agents,avoid opioid agents, Post operative nausea and vomiting prophylaxis, Patient will wear well-fitting compression stockings and receive pharmacological prophylaxis with LMWH. Encourage to mobilize out of bed after effect of general anesthesia has weaned off, Chewing gum, oral magnesium and alvimopan can be started early postoperatively, Initiation of feeding-Oral sips on day 1, step up day 2 onward, Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube, Removal of urinary catheter-after weaning from the effect of general anesthesia and drain removal -anytime within 24 hours;drain will not be removed if fluid is bilious or pus.
  Interventions: Combination Product: ERAS protocols; Combination Product: Early oral feeding; Combination Product: Prophylaxis against DVT

INTERVENTIONS:
Combination Product: ERAS protocols — ERAS protocols including avoidance of prolonged pre-operative fasting and early removal of Ryle, surgical drains and urinary catheter
  Other Names: Fast-track surgery protocols
  Groups: ERAS
Combination Product: Early oral feeding — Chewing gum, oral magnesium and alvimopan can be started early postoperatively, Initiation of feeding-Oral sips on day 1, step up day 2 onward
  Groups: ERAS
Combination Product: Prophylaxis against DVT — Patient will wear well-fitting compression stockings and receive pharmacological prophylaxis with LMWH. Encourage to mobilize out of bed after effect of general anesthesia has weaned off.
  Groups: ERAS

SUMMARY:
Although the ERAS program is widely used in elective procedures in many surgical subspecialties, the place of this program in emergency surgery remains uncertain probably because of the significant challenges in applying all ERAS pathways in the emergency setting. Nevertheless, the ERAS program is often modified in elective procedures on an individual and/ or institutional basis and thus may also have a role in the emergency setting albeit in a modified form.

DETAILED DESCRIPTION:
The cases will be randomized simply into two groups, Group (A) for conventional care and Group (B) for ERAS. Random assignment of intervention will be done after subjects have been assessed for eligibility and recruited. The sealed envelope method will be used for randomization.

Both groups will have pre-operative ryle inserted, urinary catheter applied, Tracheal intubation and with General anesthesia, exploration laparotomy Group (A) Fatsing for at least 6 hours pre-operative, No restriction of IV fluids and traditional analgesia including opiates. Post-operative Ambulation-as per patients' own request, Removal of urinary catheter when patient ambulates, patient will keep fasting for 3 days postoperative, oral fluids for 3 days, semi-solid for another 3 days and then can take full diet, removal of nasogastric tube just before starting oral fluids, drain removal just before discharge.

Group (B) Preoperative information, education and counselling, If possible, Clear fluids are allowed up to 2 h and solids up to 6 h prior to induction of anaesthesia, Short acting anesthetic agents,avoid opioid agents, Post operative nausea and vomiting prophylaxis, Patient will wear well-fitting compression stockings and receive pharmacological prophylaxis with LMWH. Encourage to mobilize out of bed after effect of general anesthesia has weaned off, Chewing gum, oral magnesium and alvimopan can be started early postoperatively, Initiation of feeding-Oral sips on day 1, step up day 2 onward, Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube, Removal of urinary catheter-after weaning from the effect of general anesthesia and drain removal -anytime within 24 hours;drain will not be removed if fluid is bilious or pus.

ELIGIBILITY:
Inclusion Criteria:

* Pateint presented with acute abdomen necessitating urgent GIT surgery

Exclusion Criteria:

* Known Chronic kidney disease/ Chronic liver disease patients Patients with history of chronic steroid abuse. Patient requiring Positive Pressure Ventilator support post operatively for more than 12 hours.

Patient presented with Acute Appendicitis or Acute Cholecystitis. Patient refusing for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented with acute abdomen or surgical peritonitis that require urgent abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to one month
  In days

SECONDARY OUTCOMES:
Time to ambulation | Up to one month
  in hours
Time to first flatus | Up to one month
  In hours
Time to first fluid diet | Up to one month
  In hours
Time to removal of drains | Up to one month
  In hours

CONTACTS AND LOCATIONS:
Overall Officials: Abd Allah Badawy, MD, Study Director — Prof. Dr.; Ashraf A Helmy, MD, Study Chair — Prof. Dr.; Ahmed A Abd ElMotleb, MD, Study Chair — Dr.

IPD SHARING:
Plan to Share IPD: Yes
After completion of study
Supporting Information: Study Protocol, CSR
Time Frame: By April 2022

REFERENCES:
- [Background] Andrews EJ, McCourt M, O'Riordain MG. Enhanced recovery after elective colorectal surgery: now the standard of care. Ir J Med Sci. 2011 Sep;180(3):633-5. doi: 10.1007/s11845-011-0709-1. Epub 2011 Apr 13. PMID 21487688
- [Background] Ansari D, Gianotti L, Schroder J, Andersson R. Fast-track surgery: procedure-specific aspects and future direction. Langenbecks Arch Surg. 2013 Jan;398(1):29-37. doi: 10.1007/s00423-012-1006-9. Epub 2012 Sep 27. PMID 23014834
- [Background] Lyon A, Payne CJ, Mackay GJ. Enhanced recovery programme in colorectal surgery: does one size fit all? World J Gastroenterol. 2012 Oct 28;18(40):5661-3. doi: 10.3748/wjg.v18.i40.5661. PMID 23155304
- [Background] Paduraru M, Ponchietti L, Casas IM, Svenningsen P, Zago M. Enhanced Recovery after Emergency Surgery: A Systematic Review. Bull Emerg Trauma. 2017 Apr;5(2):70-78. PMID 28507993
- [Result] Kehlet H, Wilmore DW. Fast-track surgery. Br J Surg. 2005 Jan;92(1):3-4. doi: 10.1002/bjs.4841. No abstract available. PMID 15635603
- [Result] ERAS Compliance Group. The Impact of Enhanced Recovery Protocol Compliance on Elective Colorectal Cancer Resection: Results From an International Registry. Ann Surg. 2015 Jun;261(6):1153-9. doi: 10.1097/SLA.0000000000001029. PMID 25671587
- [Result] Liu VX, Rosas E, Hwang J, Cain E, Foss-Durant A, Clopp M, Huang M, Lee DC, Mustille A, Kipnis P, Parodi S. Enhanced Recovery After Surgery Program Implementation in 2 Surgical Populations in an Integrated Health Care Delivery System. JAMA Surg. 2017 Jul 19;152(7):e171032. doi: 10.1001/jamasurg.2017.1032. Epub 2017 Jul 19. PMID 28492816
- [Result] Abraham N, Albayati S. Enhanced recovery after surgery programs hasten recovery after colorectal resections. World J Gastrointest Surg. 2011 Jan 27;3(1):1-6. doi: 10.4240/wjgs.v3.i1.1. PMID 21286218